CLINICAL TRIAL: NCT02870335
Title: Effectiveness of a Protocol Manual Therapy and Proprioceptive Neuromuscular Facilitation in Field Hockey Players.
Brief Title: Manual Therapy and Proprioceptive Neuromuscular Facilitation in Field Hockey Players.
Acronym: MTPNFHockeyP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID014
Record Dates: First submitted 2016-08-08; First posted 2016-08-17 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Hockey Players Whith Lower Back and Hamstring Pain
Keywords: low back; manual therapy; stretching
MeSH Terms: interventions — Musculoskeletal Manipulations; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Therapy (Experimental): The objective of treatment is to restore esta possible limitation of global mobility to major lower limb joints and remove any tensions from the musculature involved in a relevant way in this sport.
  Interventions: Other: Manual Therapy
- Proprioceptive neuromuscular facilitation (Active Comparator): It is a stretching technique with the aim of increasing the ROM. It includes passive static stretching and contract-relax.
  Interventions: Other: Proprioceptive neuromuscular facilitation

INTERVENTIONS:
Other: Manual Therapy — The patient remained lying on the gurney and the treatment was performed in the order set forth below and included: overall bilateral manipulation of L5-S1-Sacroiliac, subsequently decompression hip joint, the tibiofemoral decompression, stretching rotators hip flexion or hip and knee mobilization technique downing head and base of the fibula, tibiofibular-talus tali posteriorización decompression and with the help of a wedge to facilitate technical.
  Arms: Manual Therapy
Other: Proprioceptive neuromuscular facilitation — Stretching were conducted in the hamstrings, psoas, adductors, pyramidal, quadriceps and right above.
  Arms: Proprioceptive neuromuscular facilitation

SUMMARY:
Introduction: Field hockey is a contact sport. Semiflexion asymmetric position, along with other theories such as the weakness of the extensor muscles of the back or hamstring injury, can be causes or aggravating that suelan hockey players suffer back pain. Objectives: To observe the effectiveness of manual therapy techniques and post-isometric stretching (PNF) after three treatment sessions. In turn, know which of the two treatments have a greater benefit and longer. Methods: The population consists of grass hockey players and senior category aged between 16-30 years. They were randomly divided into two treatment groups. Group 1 corresponded to manual therapy techniques and group 2 to PNF stretching. The study duration for each subject was 5 sessions that included 3 treatment and 3 assessments. Each evaluation consisted of goniometry, balance test using the Sit and Reach, and Roland Morris questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* field hockey players (HH) (senior category).
* between 16 and 30 years.
* suffered injuries and microtraumatic not prevent them from sports.

Exclusion Criteria:

* subjects with structural abnormalities of the spine.
* plantar alterations.
* other moderate or severe musculoskeletal previous injuries in the last 6 months and prevented them make sport normally.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Dynamic balance | 6 weeks
  Was assessed using the Star Excursion Balance Test (SEBT), Which bilateral in the above (A), posteromedial (PM) and posterolateral (PL) Were used reach directions.

SECONDARY OUTCOMES:
Active Range of Moviment | 6 weeks
  Goniometry of both legs with universal goniometer external and internal rotation of the hip, hip flexion, knee flexion and ankle dorsiflexion.
Lumbar flexibility | 6 weeks
  Was assessed using the Fingertip-to-Floor Test (FFT). Subjects were placed barefoot over a 25-cm high platform, with feet together and flat, and toes on the edge pointing forward. Then, they were asked to bend the trunk from the upright position as far as possible without discomfort, while maintaining knees and arms fully extended. Flexion was held for 3 seconds and the vertical distance between the tip of the middle finger and the platform was measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Gemma Espí López, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No